CLINICAL TRIAL: NCT00473239
Title: The Pharmacokinetics of a Single Large Dose of Vitamin D3
Acronym: Stoss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: Procter and Gamble (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Creighton2
Record Dates: First submitted 2007-05-11; First posted 2007-05-15 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; cholecalciferol; 25-hydroxyvitamin D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cholecalciferol (Experimental): A single dose of 100,000 IU vitamin D
  Interventions: Drug: cholecalciferol.
- Control (No Intervention): No drug was given

INTERVENTIONS:
Drug: cholecalciferol. — 100,000 IU of Vitamin D
  Other Names: vitamin D
  Arms: cholecalciferol

SUMMARY:
When people eat a meal, some, but not all of the calcium in that meal is absorbed, that is, moved into the bloodstream. When the skin is exposed to sunlight during summer months, Vitamin D is made there and then modified into more active forms by the liver and kidneys. These more active forms of Vitamin D improve calcium absorption. Many adults living in the U.S. have little or no sun exposure and are low in Vitamin D. A single dose of 100,000 IU of Vitamin D3 has been used both as empiric treatment for Vitamin D deficiency as well as in controlled trials without risk of raising blood calcium to dangerous levels.This study is to determine the serum levels of Vitamin D and 25-hydroxyvitamin D (vitamin D after it has been modified by the liver) that can be expected when Vitamin D3 is given as a single oral dose of 100,000 IU.

DETAILED DESCRIPTION:
The group receiving the supplement will be scheduled for short visits to our research center at baseline and days 1,3,5,7 and then weekly for 3 weeks and then every other week for 6 visits (total 14 visits in 4 months). The group not receiving supplement will be scheduled for short visits at baseline and in 4 months. At the beginning of the study we will measure your height, weight, skin color, and draw blood to measure your blood levels of Vitamin D, 25-hydroxyvitamin D, calcium and parathyroid hormone. At each visit we will draw blood to measure your blood levels of Vitamin D and 25-hydroxyvitamin D. There will be fourteen blood draws for a total of 280 cc of blood drawn (about 4 teaspoons drawn each time) in the supplemented group. There will be 2 blood draws in the group not receiving supplements for a total of 60 cc of blood drawn (about 4 teaspoons drawn each time).

ELIGIBILITY:
Inclusion Criteria:

* healthy with limited sun exposure of less than 10 hours per week and daily milk consumption of less than 0.47 L (16 oz.).

Exclusion Criteria:

* those with granulomatous conditions, liver disease, kidney disease, or diabetes and those taking anticonvulsants, barbiturates, or steroids in any form.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-10; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
to assess the time course and response of serum 25-OHD with a single oral dose of 100,000 IU cholecalciferol. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Armas, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Ilahi M, Armas LA, Heaney RP. Pharmacokinetics of a single, large dose of cholecalciferol. Am J Clin Nutr. 2008 Mar;87(3):688-91. doi: 10.1093/ajcn/87.3.688. PMID 18326608